CLINICAL TRIAL: NCT01393873
Title: The Effect of Bariatric Surgery on the Progression of Diabetic Retinopathy
Brief Title: Progression of Diabetic Retinopathy Post Bariatric Surgery (BS)
Status: Terminated | Type: Observational
Why Stopped: Investigator has moved to other state.
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Heekoung A Youn, Research coordinator, NYU Langone Health
Other Study IDs: R10-02084
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Obesity; Diabetes Mellitus
Keywords: Obesity; Type 2 DM
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric surgery pts with Type 2 DM: Primary bariatric surgery pts with Type 2 DM

SUMMARY:
Studies conducted assessing diabetic eye disease have shown a progression of diabetic retinopathy with rapid improvement of glycemic control during pregnancy and in patients with type 1 diabetes. It is also well documented that bariatric surgery may result in rapid improvement of glycemic control in obese patients with type 2 diabetes. To our knowledge the progression of diabetic eye disease seen in pregnancy and type 1 diabetes has not been studied in obese type 2 diabetics undergoing bariatric surgery. To this end, this study will examine the effects of rapid glycemic control which is seen in type 2 diabetics following bariatric surgery on the progression of diabetic retinopathy.

DETAILED DESCRIPTION:
Participants will be referred from the Department of Bariatric Surgery at NYU. The investigators plan to enroll 50 patients in this pilot study.

A baseline eye exam will be conducted prior to surgery. Data, such as preoperative HbA1c level, weight, BMI, duration and control of diabetes, current medication regimen, and the grade of retinopathy will be noted. Study participants will have a baseline eye exam within three months of the scheduled surgery, followed by regular follow-up visits at 3 months, 6 months, 9 months, and 1 year. At each visit the following measures will be assessed: (1) weight, (2) blood pressure, (3) glycemic control as assessed by HbA1C, (4)level of retinopathy, and (5) visual acuity using the EDTRS acuity chart.

The eye examinations will consist of a measure of best-corrected visual acuity, slit lamp examination to assess pressure, and a dilated funduscopic examination to determine the presence and/or level of retinopathy. The level of retinopathy will be characterized as:

(0)None, (1) Mild, (2) Moderate, (3) Severe, and (4) Proliferative. In addition, the presence or absence of cystoid macular edema (CME) will be noted as (a) no CME or (b) CME present.

At the initial visit, a baseline questionnaire will be given to participants to gather background information on demographics and pertinent medical history. During each follow up visit, an additional questionnaire will be given to monitor changes in factors such as medications, blood pressure, and weight that may occur after bariatric surgery.

HbA1c measurements will be checked every 3 months in accordance with current standard of care recommendations. Due to established evidence of rapid improvement in glycemic control shortly after bariatric surgery, it is essential that the investigators have this lab data and perform funduscopic examinations at these intervals, to monitor improvement in glycemic control ascertain associations between changes in HbA1c levels and progression of retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* All patients, both male and female greater than 18 years old, with type 2 diabetes referred for bariatric surgery.

Exclusion Criteria:

* Patients will not be included in the study if they are pregnant, have HIV or any retinal vascular diseases (e.g. BRVO, CRVO) besides retinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes in the bariatric service awaiting metabolic surgery for weight reduction/glucose control therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
rapid changes in the level of retinopathy | 12 months
  whether rapid changes in the level of retinopathy do or do not occur in the transition period following surgery, where weight loss may be rapid causing improvement in insulin resistance and glycemic control.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Danoff, M.D., Principal Investigator — NYU SOM
Locations (1):
- NYU SOM, New York, New York, United States